CLINICAL TRIAL: NCT00255749
Title: Assessment of Early and Standard Intervention With Procrit® (Epoetin Alfa) 120,000 Units Once Every Three Weeks (Q3W) in Patients With Cancer Receiving Chemotherapy
Brief Title: Epoetin Alfa in Treating Patients With Anemia Who Are Undergoing Chemotherapy for Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000449950; UCLA-0504038; ORTHO-PR04-27-018
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Anemia; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: adult acute lymphoblastic leukemia in remission; progressive hairy cell leukemia, initial treatment; stage 0 chronic lymphocytic leukemia; anemia; extramedullary plasmacytoma; isolated plasmacytoma of bone; refractory multiple myeloma; monoclonal gammopathy of undetermined significance; primary systemic amyloidosis; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult T-cell leukemia/lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III mycosis fungoides/Sezary syndrome; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV mycosis fungoides/Sezary syndrome; stage IV small lymphocytic lymphoma; Waldenström macroglobulinemia; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; post-transplant lymphoproliferative disorder; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult Hodgkin lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult T-cell leukemia/lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage II adult Hodgkin lymphoma; stage II adult T-cell leukemia/lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory hairy cell leukemia; prolymphocytic leukemia; unspecified adult solid tumor, protocol specific; T-cell large granular lymphocyte leukemia
MeSH Terms: conditions — Anemia; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Precancerous Conditions; Leukemia, Lymphocytic, Chronic, B-Cell; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Waldenstrom Macroglobulinemia; Leukemia, Hairy Cell; Leukemia, Prolymphocytic; Leukemia, Large Granular Lymphocytic | interventions — Epoetin Alfa

ARMS (2):
- early intervention epoietin alfa (Experimental): Patients receive epoetin alfa subcutaneously on day 1. Treatment repeats every 21 days for up to 5 courses.
  Interventions: Biological: epoetin alfa
- standard intervention epoietin alfa (Other): Patients receive epoetin alfa as in arm I once their hemoglobin level is ≤ 10.5 g/dL.
  Interventions: Biological: epoetin alfa

INTERVENTIONS:
Biological: epoetin alfa

SUMMARY:
RATIONALE: Epoetin alfa may cause the body to make more red blood cells. It is used to treat anemia caused by cancer and chemotherapy.

PURPOSE: This randomized phase II trial is studying how well epoetin alfa works in treating patients with anemia who are undergoing chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy, in terms of maintenance of target hemoglobin and hematocrit levels, of interval dosing with epoetin alfa in patients with anemia undergoing chemotherapy for nonmyeloid cancer.
* Determine the safety of this drug in these patients.

Secondary

* Determine the quality of life of patients treated with this drug.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I (early intervention): Patients receive epoetin alfa subcutaneously on day 1. Treatment repeats every 21 days for up to 5 courses.
* Arm II (standard intervention): Patients receive epoetin alfa as in arm I once their hemoglobin level is ≤ 10.5 g/dL.

Quality of life is assessed prior to start of study treatment, at week 7 during study treatment, and after completion of study treatment.

After completion of study treatment, patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 180 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed nonmyeloid cancer

  * No history of myelodysplasia
* Baseline hemoglobin 11-12 g/dL
* No anemia due to factors other than cancer or chemotherapy (e.g., iron, cyanocobalamin [vitamin B_12], or folate deficiencies, hemolysis, or gastrointestinal bleeding)
* Receiving chemotherapy that meets the following criteria:

  * Administered weekly OR every 3 weeks
  * Must begin chemotherapy on or before the first day of study treatment
* No known, untreated CNS metastases

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent)
* Iron transferrin saturation > 20%
* No history of chronic hypercoagulable disorders (e.g., activated protein C resistance, anti-cardiolipin disorder, protein C deficiency, or protein S deficiency)

Hepatic

* Bilirubin < 2.0 mg/dL
* SGPT ≤ 3 times upper limit of normal

Renal

* Creatinine ≤ 1.5 mg/dL
* No significant, uncontrolled genitourinary disease or dysfunction

Cardiovascular

* No uncontrolled cardiac arrhythmia in the past 6 months
* No uncontrolled hypertension
* No deep vein thrombosis, ischemic stroke, or other arterial or venous thrombotic events

  * Superficial thromboses allowed
* No other significant, uncontrolled cardiovascular disease or dysfunction

Pulmonary

* No significant, uncontrolled pulmonary disease or dysfunction
* No pulmonary emboli

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No infection requiring hospitalization or antibiotics in the past 14 days
* No known hypersensitivity to mammalian cell-derived products or to human albumin
* No new onset (in the past 3 months) poorly controlled seizures
* No other active malignancy except basal cell carcinoma or carcinoma in situ
* Not an employee of the investigator or study center or family members of the employee or the investigator
* No significant, uncontrolled neurological, endocrine, or gastrointestinal disease or dysfunction

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Chemotherapy
* More than 3 months since prior erythropoietic agent (e.g., epoetin alfa, darbepoetin alfa, or gene-activated erythropoietin)
* More than 4 weeks since prior packed red blood cell transfusion
* No concurrent stem cell harvest of bone marrow
* No concurrent interleukin-11
* No other concurrent erythropoietic agent

Chemotherapy

* See Disease Characteristics
* No concurrent high-dose chemotherapy with stem cell transplantation

Radiotherapy

* No concurrent nonpalliative radiotherapy

Surgery

* More than 2 weeks since prior major surgery

Other

* At least 1 month since prior investigational agents or devices
* No concurrent high-dose IV iron supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-08; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Efficacy | 7 weeks
Safety | 7 weeks

SECONDARY OUTCOMES:
Quality of life | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John A. Glaspy, MD, MPH, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Derived] Glaspy JA, Charu V, Luo D, Moyo V, Kamin M, Wilhelm FE. Initiation of epoetin-alpha therapy at a starting dose of 120,000 units once every 3 weeks in patients with cancer receiving chemotherapy: an open-label, multicenter study with randomized and nonrandomized treatment arms. Cancer. 2009 Mar 1;115(5):1121-31. doi: 10.1002/cncr.24127. PMID 19170225